CLINICAL TRIAL: NCT03542409
Title: Assessment of Safety and Feasibility of Preoperative and Intraoperative Image-Guided Resection of Gliomas and Tumor Region-Specific Biomarker Correlation
Brief Title: Safety and Feasibility of Preoperative and Intraoperative Image-Guided Resection of Gliomas
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI77238
Record Dates: First submitted 2018-05-01; First posted 2018-05-31 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-06

CONDITIONS: Brain Tumor Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1, Group A (contrast enhancing tumor) (Experimental): Group A patients will undergo standard tumor preoperative imaging and MR perfusion scan prior to surgical resection. Group A patients will undergo standard intraoperative imaging along with MR perfusion scan during surgical resection.
  Interventions: Other: MR Perfusion Scan
- Cohort 1, Group B (non-enhancing tumor) (Experimental): Group B patients will undergo standard tumor preoperative imaging and 2HG spectroscopy scan prior to surgical resection. Group A patients will undergo standard intraoperative imaging along with 2HG spectroscopy scan during surgical resection.
  Interventions: Other: 2HG Spectroscopy Scan
- Cohort 2 (Experimental): During the analysis for cohort 1, we found significant differences in the pre MRI samples and the post intraoperative MRI samples. Cohort 2, which will include 10 additional patients, has be created to confirm these differences. Unlike cohort 1, advanced imaging (2-HG spectroscopy and MR perfusion) is not needed to make this comparison. The standard of care intraoperative MRI sequences used routinely will be sufficient for these 10 new samples. The specific aim of Cohort 2 is:
  1. Compare areas from initial surgery with that of extended resection after intraoperative SOC MRI in 10 additional subjects (Cohort 2).
  Interventions: Other: Standard of Care Intraoperative MRI

INTERVENTIONS:
Other: MR Perfusion Scan — MR perfusion scan before and during surgery.
  Arms: Cohort 1, Group A (contrast enhancing tumor)
Other: 2HG Spectroscopy Scan — 2HG spectroscopy scan before and during surgery.
  Arms: Cohort 1, Group B (non-enhancing tumor)
Other: Standard of Care Intraoperative MRI — The standard of care intraoperative MRI sequences used routinely will be sufficient for these 10 new samples.
  Arms: Cohort 2

SUMMARY:
This study evaluates the use of specialized magnetic resonance imaging (MRI) techniques including magnetic resonance (MR) perfusion and 2-hydroxyglutarate (2HG) spectroscopy in the surgical treatment of gliomas.

Cohort 1 participants will undergo an MR perfusion scan or 2-HG spectroscopy prior to surgery and intra-operatively.

Cohort 2 participants will only undergo standard of care imaging and tumor acquisition. Participant participation will end at the completion of surgery and will be transitioned to standard of care follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Suspected glioma (grade II, III, or IV)
* Preoperative MR perfusion (enhancing tumors)
* Preoperative MR 2-HG spectroscopy (nonenhancing tumors)Patient indicated for surgical resection, standard radiation, and standard chemotherapy as a standard of care
* Karnofsky performance status ≥ 60
* Life expectancy > 12 weeks
* Cohort 1: Ability to comply with study and follow-up procedures
* Cohort 2: Ability to comply with study procedures

Exclusion Criteria:

* Prior diagnosis of intracranial glioma
* Other malignancy with expected need for systemic therapy within 3 years
* Inability to have 6000 grays of radiation to the brain
* Need for urgent palliative intervention for primary disease (e.g., impending herniation)
* Evidence of bleeding diathesis or coagulopathy
* History of intracerebral abscess within 6 months prior to Day 0
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study
* Pregnant females
* Subjects unable to undergo an MRI with contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Intraoperative Imaging Completion | 1 day
  This is a feasibility study to see whether advanced imaging modalities can be used intraoperatively so the primary outcome is a yes/no regarding completion of imaging.
Incidence of Patient Complications Following Tumor Resection | 1 year
  Any surgical complications at post-op, hospital discharge, 1-month, 3-months, 6-months, and 1 year following surgery using the Common Terminology Criteria for Adverse Events (CTCAE)

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided